CLINICAL TRIAL: NCT00004082
Title: A Phase I Study of Docetaxel (Taxotere), Carboplatin, and Gemcitabine (DoCaGem) as First-Line Therapy for Patients With High-Risk Epithelial Tumors of Mullerian Origin
Brief Title: Combination Chemotherapy in Treating Patients With Previously Untreated, Newly Diagnosed Epithelial Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: BIH-99-1285; CDR0000067293 (Registry Identifier: PDQ (Physician Data Query)); NCI-V99-1566
Record Dates: First submitted 1999-12-10; First posted 2004-04-12 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2010-11

CONDITIONS: Endometrial Cancer; Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; stage III endometrial carcinoma; stage IV endometrial carcinoma; endometrial adenocarcinoma; fallopian tube cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Endometrial Neoplasms; Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Carboplatin; Docetaxel; Gemcitabine

INTERVENTIONS:
Drug: carboplatin
Drug: docetaxel
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combining docetaxel, carboplatin, and gemcitabine in treating patients who have previously untreated, newly diagnosed epithelial cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of docetaxel, carboplatin, and gemcitabine in patients with previously untreated, newly diagnosed, high-risk epithelial cancer of mullerian origin.

OUTLINE: This is a dose-escalation study of docetaxel and gemcitabine. Patients receive docetaxel IV over 30 minutes and gemcitabine IV over 30 minutes on days 1 and 8. Carboplatin IV is administered over 30 minutes on day 1. Treatment repeats every 21-28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3-5 patients receive escalating doses of docetaxel and gemcitabine until the maximum tolerated dose is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 5 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: A total of 20-30 patients will be accrued for this study within 1.5-2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed, newly diagnosed, high-risk epithelial tumors of mullerian origin, including: Ovarian epithelial cancer Peritoneal papillary serous cancer Primary fallopian tube cancer Endometrial cancer High-risk is defined as: Any amount of gross residual disease remaining at the time of initial debulking surgery AND/OR Any radiographic or physical exam evidence of disease after surgery AND/OR Disease outside of the abdomen (e.g., malignant pleural effusion) AND/OR Parenchymal liver, spleen, or lung metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: More than 2 months Hematopoietic: WBC at least 3,000/mm3 Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than upper limit of normal (ULN) Alkaline phosphatase no greater than 2.5 times ULN SGOT and SGPT no greater than 1.5 times ULN Renal: Creatinine no greater than 1.5 mg/dL Creatinine clearance at least 35 mL/min Cardiovascular: Acceptable cardiac exam No active cardiac ischemia Pulmonary: Acceptable pulmonary exam No active pulmonary infection or compromise Other: Not pregnant or nursing No peripheral neuropathy grade 2 or greater No other debilitating medical or psychiatric conditions that would preclude study No other malignancy within the past 3 years except limited stage basal or squamous cell skin cancer or carcinoma in situ of the cervix No evidence of infection Adequate bowel function, oral intake, and wound healing ability

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior cytokine therapy for epithelial tumors of mullerian origin Chemotherapy: No more than 1 prior chemotherapy regimen for epithelial tumors of mullerian origin At least 3 years since other prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior pelvic radiotherapy Surgery: See Disease Characteristics At least 7 days since prior surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-07; Primary Completion 2003-09 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen A. Cannistra, MD, Study Chair — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States